CLINICAL TRIAL: NCT07127484
Title: Efficacy and Safety of Hemoadsorption for Severe Ischemic Stroke
Brief Title: Hemoadsorption for Severe Ischemic Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Collaborators: The Second People's Hospital of Wuhu (Unknown); Anqing People's Hospital of Anhui Medical University (Unknown); Beijing Tiantan Hospital (Other); Gansu Provincial Central Hospital (Unknown); Baotou Central Hospital (Other); The NO.1 People's Hospital of Shizuishan (Unknown); Fuyang people's hospital (Other); Second People's Hospital of Hefei City (Other); The First Affiliated Hospital of Zhengzhou University (Other); Luan people's hospital (Unknown)
Responsible Party: Principal Investigator, Jie Xu, Director, First Affiliated Hospital of Wannan Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202510
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke; Hemoadsorption
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard treatment group (No Intervention)
- standard treatment plus hemoadsorption group (Other)
  Interventions: Procedure: Hemoadsorption

INTERVENTIONS:
Procedure: Hemoadsorption — Patients in intervention group will receive standard treatment plus hemoadsorption therapy administered once on days 1, 3, and 5 following enrollment.
  Arms: standard treatment plus hemoadsorption group

SUMMARY:
This is a multicenter, randomized-controlled, open-label, blinded endpoint clinical trial that aims to evaluate the efficacy and safety of hemoadsorption for severe ischemic stroke

DETAILED DESCRIPTION:
This is a multicenter, randomized-controlled, open-label, blinded endpoint clinical trial that aims to evaluate the efficacy and safety of hemoadsorption for severe ischemic stroke. During the study period, a total of 116 patients with severe ischemic stroke will be enrolled from 10 centers. To evaluate whether adjunctive hemoadsorption therapy combined with standard treatment can reduce the incidence of severe adverse functional outcomes (modified Rankin Scale [mRS] 4-6) at 90 days. Patients in control group will receive standard treatment, and those in the other group will receive standard treatment plus hemoadsorption therapy administered once on days 1, 3, and 5 following enrollment. Study visits will be performed on the day of randomization, at treatment period, at day 7, at day 14 or hospital discharge and at day 90. In addition to the primary endpoint, the study will evaluate whether hemoadsorption can reduce acute-phase inflammatory cytokine levels and decrease the incidence of complications including hemorrhagic transformation, malignant cerebral edema, and pulmonary infections in severe ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1.18 years ≤ age < 80 years; 2.Pre-stroke mRS score ≤ 1; 3.Anterior circulation cerebral infarction within 48 hours of onset, meeting at least one of the following:

1. 15≤ NIHSS score ≤32;
2. 3<GCS score ≤12;
3. CT hypodensity area >1/2 of the MCA territory; 4.hs-CRP ≥2 mg/L at randomization; 5.If reperfusion therapy is performed, no improvement in NIHSS score (still ≤32) post-treatment; 6.Signed informed consent obtained.

Exclusion Criteria:

1. Hemorrhagic transformation of PH2 type prior to randomization;
2. Brain herniation or decompressive craniectomy performed before randomization;
3. Hemodynamic instability refractory to medical correction (systolic blood pressure <70 mmHg or diastolic blood pressure <50 mmHg) or decompensated heart failure (NYHA Class III or IV);
4. Severe hepatic impairment (defined as ALT >2 times the upper limit of normal or AST >2 times the upper limit of normal) and renal impairment (defined as serum creatinine >1.5 times the upper limit of normal or estimated glomerular filtration rate [eGFR] <50 mL/min);
5. Coagulopathy or thrombocytopenia (platelet count <100×10⁹/L);
6. Deep vein thrombosis (DVT) of the lower extremities before randomization;
7. Life expectancy <90 days due to malignancy;
8. Participation in another drug or device clinical trial within the past 30 days or ongoing enrollment in such trials;
9. Women of childbearing potential with a negative pregnancy test who refuse to use effective contraception, or pregnant/lactating women;
10. Absolute contraindications to hemoadsorption therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of severe adverse functional outcomes (modified Rankin Scale [mRS] 4-6) | From enrollment to the end of treatment at 90 days